CLINICAL TRIAL: NCT03460704
Title: Efficacy and Safety of 12 Months of Therapy With Inhaled Colistimethate Sodium in Subjects With Non-cystic Fibrosis Bronchiectasis Chronically Infected With P. Aeruginosa
Brief Title: Trial in Non-cystic Fibrosis Bronchiectasis Patients With Chronic Lung Infections Treated With Colistimethate Sodium.
Acronym: PROMIS-II
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was brought to an early close in March 2022 due to major ongoing recruitment issues primarily related to the COVID-19 pandemic and concerns regarding the continued randomization and exposure of subjects to placebo in the study.
Sponsor: Zambon SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Z7224L02; 2016-004558-13 (EudraCT Number)
Record Dates: First submitted 2018-02-14; First posted 2018-03-09 (Actual); Results first posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Non Cystic Fibrosis Bronchiectasis
Keywords: NCFB; NCFB pulmonary exacerbation; Bronchiectasis
MeSH Terms: conditions — Bronchiectasis | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CMS (Colistimethate Sodium) (Experimental): Inhaled colistimethate sodium twice daily. The active pharmaceutical ingredient consisting of pure CMS one million international units (MIU) / 80 mg of CMS / 33 mg colistin base activity (CBA) was provided as a powder for nebuliser solution in 10R Internation Organization for Standardization (ISO) glass vials.
  Interventions: Drug: CMS
- Placebo (Placebo Comparator): Saline solution inhaled twice daily, provided and administered at the same way of the IMP.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CMS — 1 MIU equivalent to 80 mg colistimethate sodium diluted in 1 mL saline solution 0.45%. Investigational Medicinal Product (IMP) glass vials were shrink wrapped in opaque white plastic and provided in boxes of 30 vials (two weeks of b.i.d. dosing).
  The 1 MIU/ml CMS/0.45% saline solution was transferred from the glass vial into a specific nebuliser system fitted with a 0.3 mL medication chamber, for administration by inhalation. This delivered a nominal dose of 0.3 MIU/24 mg CMS (11 mg CBA) from the device.
  The first dose of the IMP was administered at the site under the supervision of the site staff and subjects were instructed how to prepare and self-administer the IMP at home via a specific nebuliser system, b.i.d. (morning and evening) over aperiod of 12 month.
  At least 10 minutes (min) before each administration, an inhaled short-acting bronchodilator (e.g. salbutamol/albuterol), supplied by the Sponsor, could be taken to improve tolerability.
  Other Names: Promixin
  Arms: CMS (Colistimethate Sodium)
Other: Placebo — 1 mL saline solution 0.45%. The placebo was made up of identical empty glass vials to which the same saline solution diluent was added in exactly the same way as the reconstitution of the active treatment by injecting the diluent through the rubber stopper. The glass vials were shrink wrapped with opaque white plastic to mantain the blind.
  Other Names: Saline Solution
  Arms: Placebo

SUMMARY:
The primary objective of the trial was to investigate the effect of the use of inhaled colistimethate sodium (CMS), administered twice a day (b.i.d.) via a specific nebulizer for 12 months, compared to placebo in subjects with non-cystic fibrosis bronchiectasis (NCFB) chronically infected with P. aeruginosa on the annualised frequency of pulmonary exacerbations.

DETAILED DESCRIPTION:
This was a randomised, multi-centre, double-blind, placebo-controlled, parallel-group interventional trial in subjects with NCFB chronic P. aeruginosa infection. Subjects were randomised to CMS or placebo in a 1:1 ratio. The study consisted of 7 clinic visits with a follow-up phone call 12.5 month after randomisation or 2 weeks after discontinuation of treatment. Additional clinic visits, where feasible, and weekly phone calls were conducted during or after pulmonary exacerbations (or any episodes of pneumonia) until resolution.

Every effort was made to have all planned and unscheduled visits at the study site. Mandatory on-site visits were Screening Visit (Visit 1) and Randomisation (Visit 2). However, if one of the visits after Visit 2 could not be performed at site due to COVID-19, remote visits (e.g., by telephone) were permitted. If the final visit (Visit 7) had to be conducted remotely, the subjects were asked to return to the clinic for on-site assessments at the earliest opportunity.

After consulting with the US Food and Drug Administration, the study was brought to an early close primarily due to the difficulty of recruiting subjects in the context of the COVID pandemic, but also due to the potential for loss of scientific equipoise and the ethical implications of continuing to expose subjects to placebo given the positive results from PROMIS I. Recruitment to PROMIS II was stopped as of 27 October 2021, with the study terminated as of 15 March 2022. The study was not stopped prematurely due to any safety or futility concerns and the accrued data were fully analysed and are presented.

ELIGIBILITY:
Inclusion Criteria:

1. are able and willing to give informed consent, following a detailed explanation of partecipation in the protocol and signed consent obtained;
2. aged 18 years or older of either gender;
3. diagnosed with NCFB by computerised tomography (CT) or high-resolution CT(HRCT) as recorded in the subject's notes and this is their predominant condition being treated;
4. had at least 2 NCFB pulmonary exacerbations requiring oral or inhaled antibiotics or 1 NCFB pulmonary exacerbation requiring intravenous antibiotics in the 12 months preceding the Screening Visit (Visit 1) and had no pulmonary exacerbation with or without treatment during the period between Visit 1 and Visit 2;
5. have a documented history of P. aeruginosa infection;
6. are clinically stable and have not required a change in pulmonary treatment for at least 30 days before the Screening Visit (Visit 1);
7. have pre-bronchodilator FEV1 ≥25% of predicted;
8. had a positive sputum culture for P. aeruginosa from an adequate sample taken at the Screening Visit (Visit 1) or during the screening period.

Exclusion Criteria:

1. known bronchiectasis as a consequence of cystic fibrosis (CF);
2. known history of hypogammaglobulinaemia requiring treatment with immunoglobulin, unless fully replaced and considered immuno-competent by the Investigator;
3. myasthenia gravis or porphyria;
4. severe cardiovascular disease such as severe uncontrolled hypertension, ischaemic heart disease or cardiac arrhythmia and any other conditions that would confound the evaluation of safety, in the opinion of the Investigator;
5. had major surgery in the 3 months prior to the Screening Visit (Visit 1) or planned inpatient major surgery during the study period;
6. receiving treatment for allergic bronchopulmonary aspergillosis (ABPA);
7. massive haemoptysis (greater than or equal to 300 mL or requiring blood transfusion) in the preceding 4 weeks before Screening Visit (Visit 1) or between Visit 1 and Visit 2;
8. respiratory failure that would compromise patient safety or confound the evaluation of safety or efficacy of the study in the opinion of the Investigator;
9. current active malignancy, except for basal cell carcinoma or squamous cell carcinoma of the skin without metastases;
10. taking immunosuppressive medications (such as azathioprine, cyclosporine, tacrolimus, sirolimus, mycophenolate, rituximab), and/or anti cytokine medications (such as anti-IL-6 and anti-tumour alpha necrosis factor products) in the preceding year before the Screening Visit (Visit 1);
11. known history of human immunodeficiency virus (HIV);
12. current treatment for non-tuberculous mycobacterial (NTM) lung disease or tuberculosis;
13. known or suspected to be allergic or unable to tolerate colistimethate sodium (intravenous or inhaled) or other polymixins, including evidence of bronchial hyper-reactivity following inhaled colistimethate sodium;
14. treatment with long term (≥ 30 days) prednisone at a dose of greater than 15 mg a day (or equivalent dose of any other corticosteroid) started within six months of the Screening Visit (Visit 1);
15. new maintenance treatment with any oral macrolides ( (e.g. azithromycin/erythromycin/clarithromycin) within 30 days of the Screening Visit (Visit 1) or started between Visit 1 and Visit 2;
16. use of any intravenous or intramuscular or oral or inhaled anti-pseudomonal antibiotic (except chronic macrolides with a stable dose) within 30 days prior to the Screening Visit (Visit 1) and between Visit 1 and Visit 2;
17. pregnant or breast feeding or plan to become pregnant over the next two years or of child- bearing potential and unwilling to use a reliable method of contraception for at least one month before randomisation and throughout their involvement in the trial;
18. significant abnormality in clinical evaluations and/or laboratory tests (physical examination, vital signs, haematology, clinical chemistry, clinically relevant impaired renal function, defined as serum creatinine levels ≥2.0x upper limit of normal, ECG) endangering the safe participation of the patient in the study at the Screening Visit (Visit 1) and during the study;
19. participated in another investigational, interventional trial within 30 days prior to the Screening Visit (Visit 1);
20. in the opinion of the Investigator not suitable for inclusion for whatever reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paola Castellani, MD, Principal Investigator — Zambon S.p.A.
Locations (83):
- United States (27):
  - Zambon Investigative Site, Newport Beach, California
  - Zambon Investigative Site, Palm Springs, California
  - Zambon Investigative Site, Reseda, California
  - Zambon investigative site, San Diego, California
  - Zambon Investgative Site, San Diego, California
  - Zambon Investigative Site, Centennial, Colorado
  - Zambon Investigative Site, Jacksonville, Florida
  - Zambon Investigative Site, Kissimmee, Florida
  - Zambon Investigative Site, Orlando, Florida
  - Zambon investigative Site, St. Petersburg, Florida
  - Zambon Investigative Site, St. Petersburg, Florida
  - Zambon Investigative Site, Weston, Florida
  - Zambon Investigative Site, Chicago, Illinois
  - Zambon Investigative Site, Michigan City, Indiana
  - Zambon Investigative Site, Louisville, Kentucky
  - Zambon Investigative Site, Rochester, Minnesota
  - Zambon Investigative Site, Chesterfield, Missouri
  - Zambon Investigative Site, Lebanon, New Hampshire
  - Zambon Investigative Site, New York, New York
  - Zambon investigative site, Chapel Hill, North Carolina
  - Zambon Investigative Site, Durham, North Carolina
  - Zambon investigative site, Winston-Salem, North Carolina
  - Zambon Investigative Site, Portland, Oregon
  - Zambon Investigative Site, Tyler, Texas
  - ZambonInvestigative Site, Abingdon, Virginia
  - Zambon investigative site, Richmond, Virginia
  - Zambon Investigative Site, Northwest, Washington
- Argentina (5):
  - Zambon Investigative Site, Buenos Aires
  - Zambon investigative site, Buenos Aires
  - Zambon Investigative Site, Quilmes
  - Zambon Investigative Site, San Miguel de Tucumán
  - Zambon Investigative Site, Santa Fe
- Australia (6):
  - Zambon Investigative Site, Adelaide
  - Zambon investigative site, Concord
  - Zambon investigative site, Greenslopes
  - Zambon Investigative Site, Kent Town
  - Zambon Investigative Site, South Brisbane
  - Zambon investigative site, Spearwood
- Canada (7):
  - Zambon investigative Site, Burlington
  - Zambon investigative site, Kelowna
  - Zambon Investigative Site, London
  - Zambon Investigative Site, Montreal
  - Zambon Investigative Site, Ottawa
  - Zambon Investigative Site, Québec
  - Zambon Investigative Site, Winnipeg
- France (10):
  - Zambon Investigative Site, Amiens
  - Zambon investigative site, Brest
  - Zambon Investigative Site, Créteil
  - Zambon investigative site, La Tronche
  - Zambon investigative site, Lyon
  - Zambon Investigative Site, Montpellier
  - Zambon investigative site, Nice
  - Zambon Investigative Site, Pessac
  - Zambon investigative site, Reims
  - Zambon Investigative Site, Toulouse
- Germany (2):
  - Zambon Investigative Site, Frankfurt
  - Zambon Investigative Site, Hanover
- Zambon Investigative Site, Athens, Greece
- Israel (3):
  - Zambon Investigative Site, Haifa
  - Zambon Investigative Site, Jerusalem
  - Zambon Investigative Site, Kfar Saba
- Italy (2):
  - Zambon Investigative Site, Milan
  - Zambon Investigative Site, Monza
- New Zealand (4):
  - Zambon Investigative Site, Christchurch
  - Zambon Investigative Site, Havelock North
  - Zambon Investigative Site, Mount Cook
  - Zambon Investigative Site, Tauranga
- Poland (14):
  - Zambon Investigative Site, Bialystok
  - Zambon Investigative Site, Bielsko-Biala
  - Zambon Investigative Site, Grudziądz
  - Zambon Investigative Site, Krakow
  - Zambon Investigative Site, Legnica
  - Zambon Investigative Site, Lodz
  - Zambon Investigative Site, Lublin
  - Zambon Investigative Site, Ostrowiec Świętokrzyski
  - Zambon Investigative Site, Piaseczno
  - Zambon Investigative Site, Proszowice
  - Zambon Investigative Site, Rzeszów
  - Zambon Investigative Site, Sosnowiec
  - Zambon Investigative Site, Warsaw
  - Zambon Investigative Site, Wroclaw
- Portugal (2):
  - Zambon Investigative Site, Guimarães
  - Zambon Investigative Site, Lisbon

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was halted with 287 subjects randomised.
Groups:
- CMS (Colistimethate Sodium): Inhaled colistimethate sodium twice daily. The active pharmaceutical ingredient consisting of pure CMS one million international units (MIU) / 80 mg of CMS / 33 mg colistin base activity (CBA) was provided as a powder for nebuliser solution in 10R Internation Organization for Standardization (ISO) glass vials.
  CMS: 1 MIU equivalent to 80 mg colistimethate sodium diluted in 1 mL saline solution 0.45%. Investigational Medicinal Product (IMP) glass vials were shrink wrapped in opaque white plastic and provided in boxes of 30 vials (two weeks of b.i.d. dosing).
  The 1 MIU/ml CMS/0.45% saline solution was transferred from the glass vial into a specific nebuliser system fitted with a 0.3 mL medication chamber, for administration by inhalation. This delivered a nominal dose of 0.3 MIU/24 mg CMS (11 mg CBA) from the device.
  The first dose of the IMP was administered at the site under the supervision of the site staff and subjects were instructed how to prepare and self-administer the IMP at home via a specific nebuliser system, b.i.d. (morning and evening) over aperiod of 12 month.
  At least 10 minutes (min) before each administration, an inhaled short-acting bronchodilator (e.g. salbutamol/albuterol), supplied by the Sponsor, could be taken to improve tolerability.
Period: Overall Study
Arm/Group | CMS (Colistimethate Sodium) | Placebo
Started | 152 | 135
Modified Intention to Treat Population - (mITT) | 152 | 135
Safety Population - (SAF) | 152 | 135
Per-Protocol Population - (PP) | 112 | 98
Completed | 94 | 89
Not Completed | 58 | 46
Not completed — Withdrawal by Subject | 11 | 14
Not completed — Study terminated by the Sponsor | 29 | 19
Not completed — Adverse Event | 10 | 5
Not completed — Death | 3 | 2
Not completed — Non-Compliance with Study Drug | 3 | 0
Not completed — Protocol-Specified Withdrawal Criterion Met | 0 | 5
Not completed — Other | 2 | 1

BASELINE CHARACTERISTICS:
Population: The modified Intention-To-Treat (mITT) Population is the Full Analysis Set and comprised all subjects who provided informed consent, were randomised and received at least 1 dose or partial dose of the IMP.
Groups:
- Total: Total of all reporting groups
Arm/Group | CMS (Colistimethate Sodium) | Placebo | Total
Number analyzed (Participants) | 152 | 135 | 287
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 85 | 73 | 158
  >=65 years | 67 | 62 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (15.19) | 59.6 (14.73) | 59.7 (14.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 94 | 198
  Male | 48 | 41 | 89
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 146 | 130 | 276
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Greece | 2 | 1 | 3
  New Zealand | 4 | 2 | 6
  Canada | 9 | 10 | 19
  Argentina | 56 | 52 | 108
  United States | 30 | 20 | 50
  Poland | 22 | 26 | 48
  Italy | 1 | 0 | 1
  Israel | 1 | 3 | 4
  Australia | 7 | 6 | 13
  France | 18 | 12 | 30
  Portugal | 1 | 1 | 2
  Germany | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Mean Annual Non-cystic Fibrosis Bronchiectasis (NCFB) Pulmonary Exacerbation Rate
Description: The primary efficacy assessment for an individual subject was the frequency of pulmonary exacerbations (exacerbation rate). A pulmonary exacerbation was defined as the presence concurrently of at least three of the following eight symptoms/signs for at least 24 hours:
  * increased cough;
  * increased sputum volume and/or consistency;
  * increased sputum purulence;
  * new or increased haemoptysis;
  * increased wheezing;
  * increased dyspnoea;
  * increased fatigue/malaise and
  * episodes of fever (temperature ≥38°C). AND It was clinically determined that the subject required and was prescribed systemic antibiotic therapy. AND The episode of exacerbation lasted for at least 24 hours. The overall episode of exacerbation needs to last at least 24 hours, but individual symptoms/signs can last less than 24 hours (e.g, a temperature)
Time Frame: 12 months
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: Number of Pulmonary Exacerbations
Arm/Group | CMS (Colistimethate Sodium) | Placebo
Number analyzed (Participants) | 152 | 135
Number of Pulmonary Exacerbations | 0.889 [0.722 to 1.093] | 0.885 [0.710 to 1.103]
Statistical Analysis 1: Comparison: CMS (Colistimethate Sodium) vs Placebo; The number of NCFB pulmonary exacerbations was compared between treatment groups using a negative binomial model including treatment, country, and baseline use of stable concomitant therapy with oral macrolides as fixed effects and log-exposure time on treatment as an offset; Test type: Superiority; p = 0.97889, negative binomial model; LS Mean rate ratio = 1.004, 95% CI 2-sided [0.747 to 1.349]

ADVERSE EVENTS:
Time Frame: All AEs occurring from Visit 2 (day 0 = first IMP administration) until the follow-up phone call (2 weeks +/- 3 days after the end of treatment = totally up to 54 weeks +/- 3 days from the study Day 0.
Description: An AE is "any untoward medical occurrence in a patient or clinical trial subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment". An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an IMP, whether or not considered related to the IMP.
Groups:
- CMS (Colistimethate Sodium) (SAF): Inhaled colistimethate sodium twice daily. The active pharmaceutical ingredient consisting of pure CMS one million international units (MIU) / 80 mg of CMS / 33 mg colistin base activity (CBA) was provided as a powder for nebuliser solution in 10R Internation Organization for Standardization (ISO) glass vials.
  CMS: 1 MIU equivalent to 80 mg colistimethate sodium diluted in 1 mL saline solution 0.45%. Investigational Medicinal Product (IMP) glass vials were shrink wrapped in opaque white plastic and provided in boxes of 30 vials (two weeks of b.i.d. dosing).
  The 1 MIU/ml CMS/0.45% saline solution was transferred from the glass vial into a specific nebuliser system fitted with a 0.3 mL medication chamber, for administration by inhalation. This delivered a nominal dose of 0.3 MIU/24 mg CMS (11 mg CBA) from the device.
  The first dose of the IMP was administered at the site under the supervision of the site staff and subjects were instructed how to prepare and self-administer the IMP at home via a specific nebuliser system, b.i.d. (morning and evening) over aperiod of 12 month.
  At least 10 minutes (min) before each administration, an inhaled short-acting bronchodilator (e.g. salbutamol/albuterol), supplied by the Sponsor, could be taken to improve tolerability.
- Placebo (SAF): Saline solution inhaled twice daily, provided and administered at the same way of the IMP.
  Placebo: 1 mL saline solution 0.45%. The placebo was made up of identical empty glass vials to which the same saline solution diluent was added in exactly the same way as the reconstitution of the active treatment by injecting the diluent through the rubber stopper. The glass vials were shrink wrapped with opaque white plastic to mantain the blind.
Arm/Group | CMS (Colistimethate Sodium) (SAF) | Placebo (SAF)
All-Cause Mortality (participants affected / at risk) | 3/152 | 2/135
Serious Adverse Events (participants affected / at risk) | 27/152 | 17/135
Other Adverse Events (participants affected / at risk) | 123/152 | 104/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CMS (Colistimethate Sodium) (SAF) (N=152) | Placebo (SAF) (N=135)
Infective exacerbation of bronchiectasis (Infections and infestations) | 12 (12) | 10 (11)
COVID-19 (Infections and infestations) | 3 (3) | 0 (0)
Brain abscess (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pseudomonas infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Adams-Stokes syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Sinus arrest (Cardiac disorders) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CMS (Colistimethate Sodium) (SAF) (N=152) | Placebo (SAF) (N=135)
Asthma (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (3)
Constipation (Gastrointestinal disorders) | 4 (5) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 3 (4)
Muscoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 3 (3)
Pyrexia (General disorders) | 1 (1) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Syncope (Nervous system disorders) | 3 (3) | 0 (0)
Exposure to contaminated device (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Weight decreased (Investigations) | 0 (0) | 3 (3)
Chronic sinusitis (Infections and infestations) | 3 (6) | 0 (0)
Infective exacerbation of bronchiectasis (Infections and infestations) | 69 (111) | 67 (103)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (15) | 9 (10)
Headache (Nervous system disorders) | 7 (7) | 8 (8)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 9 (15) | 5 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 6 (7)
COVID-19 (Infections and infestations) | 8 (8) | 4 (4)
Sinusitis (Infections and infestations) | 6 (7) | 6 (10)
Diarrhoea (Gastrointestinal disorders) | 5 (8) | 6 (7)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 3 (7)
Nasopharyngitis (Infections and infestations) | 2 (2) | 6 (6)
Fatigue (General disorders) | 6 (7) | 2 (2)
Hypertension (Vascular disorders) | 3 (3) | 4 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Influenza (Infections and infestations) | 4 (4) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 3 (4) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-07-22): https://cdn.clinicaltrials.gov/large-docs/04/NCT03460704/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-08): https://cdn.clinicaltrials.gov/large-docs/04/NCT03460704/SAP_001.pdf